CLINICAL TRIAL: NCT07091448
Title: Prospective, Assessment of Alveolar Ridge Preservation Using Biotivity™ Amnion Chorion Membranein Atraumatic Extraction Socket
Brief Title: Biotivity A-C Membrane Socket Preservation Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00114841
Record Dates: First submitted 2025-06-24; First posted 2025-07-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alveolar Ridge Preservation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Alveolar ridge preservation with amnion chorion membrane (Experimental): The patients in both groups will go through the same treatment but with two different barrier membrane depending on the assigned group. The patients in this group will have alveolar ridge preservation with the amnion chorion membrane called Biotivity™ A-C Plus.
  Interventions: Device: Amnion chorion membrane
- Alveolar ridge preservation with collagen membrane (Active Comparator): The patients in both groups will go through the same treatment but with two different barrier membrane depending on the assigned group. The patients in this group will have alveolar ridge preservation with the amnion chorion membrane called CopiOs.
  Interventions: Device: Collagen membrane

INTERVENTIONS:
Device: Amnion chorion membrane — Alveolar ridge preservation of a single extraction socket site with a barrier membrane Biotivity™ A/C Plus.
  Arms: Alveolar ridge preservation with amnion chorion membrane
Device: Collagen membrane — Alveolar ridge preservation of a single extraction socket site with a barrier membrane CopiOs..
  Arms: Alveolar ridge preservation with collagen membrane

SUMMARY:
This is a prospective, randomized controlled pilot clinical trial evaluating the efficacy of a human placental-derived amnion chorion membrane (Biotivity™ A/C Plus Membrane) versus a conventional collagen membrane in alveolar ridge preservation (ARP) following atraumatic extraction of single posterior teeth. A total of 12 subjects will be enrolled at the University of Maryland School of Dentistry. The study aims to assess both soft tissue wound healing and hard/soft tissue dimensional changes over a 5-month period prior to dental implant placement.

Throughout the approximately 6-month study duration, participants will undergo oral exams, x-rays, surgical procedures, and follow-up visits. All participants will undergo routine tooth extraction, bone graft material and barrier placement, and dental implant placement.

Participation in the study is voluntary, and the alternative is to continue routine dental care. Risks include minor discomfort from procedures such as tooth extraction and implant placement. The major benefit of participation in the study is the preservation of jaw dimensions following extraction, which will simplify the placement of a dental implant.

DETAILED DESCRIPTION:
This randomized, controlled, parallel-arm clinical study investigates the use of Biotivity™ A/C Plus Membrane, a bioactive human amnion chorion-derived barrier membrane, in alveolar ridge preservation (ARP) of Type I or II extraction sockets. Subjects will be randomized to receive either the investigational amnion chorion membrane or a conventional collagen membrane (CopiOs Extend) over cancellous allograft (Puros®) after flapless tooth extraction in the premolar or molar region (excluding third molars).

The study will evaluate:

Primary outcome: soft tissue wound healing over 5 months using standardized wound healing indices.

Secondary outcomes: hard and soft tissue dimensional changes using CBCT and intraoral scanning, histologic evaluation of new bone formation, and implant placement feasibility.

Subjects will be followed across nine visits, including baseline (screening), ARP surgery, post-operative evaluations at multiple time points, and re-entry for implant placement at 5 months. The final implant-supported restoration will be delivered after implant integration, with continued follow-up for histologic and radiographic outcomes.

This study aims to determine whether the amnion chorion membrane provides superior soft tissue healing and volumetric bone preservation compared to conventional membranes in ARP procedures, with the goal of improving clinical outcomes in implant dentistry.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. At least 18 years old
3. In need of one posterior tooth (premolar or molar), excluding third molars, planned for extraction and replacement with a dental implant
4. Type I or II extraction socket/ ridge identified at the time of enrolment with cone-beam CT scan
5. At least one retained natural tooth adjacent to the study site

Exclusion criteria

1. Insufficient interocclusal or interdental space to allow for an implant- supported prosthesis
2. Previous interventions performed involving soft and/or bone grafting in the study site
3. Active caries
4. Uncontrolled periodontal disease present
5. Evidence of active periapical, radicular, or endodontic lesions on teeth adjacent to study site
6. History of recent extraction of an adjacent tooth (mesial and distal) to study site within 6 months of enrollment
7. Current smoker with self-reported history of more than 10 cigarettes or equivalent per day
8. Self-reported use of smokeless tobacco or e-cigarette
9. Self-reported history of current alcohol or drug abuse
10. Systemic or local disease or condition that would compromise bone metabolism, post-operative healing and/or osseointegration e.g. uncontrolled diabetes with self-reported most recent HbA1c > 8.0 within last six-month13,14
11. Systemic corticosteroids or any other medication that would influence bone metabolism, post-operative healing, and/or osseointegration
12. Pregnancy, as confirmed by a urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Soft Tissue Wound Healing Score Using Wound Healing Indices | Over the course of the study (From the time of study enrollment Alveolar Ridge Preservation [Visit 2] to 5-month dental implant placement [Visit6].
  Wound healing will be assessed during post-surgery follow-up visits using the Early Wound Healing Index (Wachtel et al., 2003), which classifies flap closure into five categories (1 = complete closure, no fibrin; 5 = necrosis), and Wound Healing Index (WHI) described by Huang (2025 ) with three categories (1 = uneventful healing with no gingival edema, erythema, suppuration, patient dis-comfort, or ﬂap dehiscence; 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or ﬂap dehiscence, but no suppuration; 3 = poor wound healing with signiﬁcant gingival edema, erythema, patient discomfort, ﬂap dehiscence, or any suppuration.) Scores will be assigned by a blinded examiner. Data will be reported as the number of participants per score category and the median EHI score per treatment group.

SECONDARY OUTCOMES:
Radiographic measurement of Mean Change at 4 Months Measured by CBCT | Over the course of the study (4 months, From the time of study enrollment Alveolar Ridge Preservation [Visit 2] to 6-month dental implant placement [Visit 9]).
  Vertical and volumetric changes in alveolar ridge dimensions will be assessed using cone-beam computed tomography (CBCT) taken at baseline (post-extraction) and 4 months after alveolar ridge preservation.
  Vertical bone height will be measured at the mid-buccal point from the cementoenamel junction (CEJ) to the alveolar crest.
  Volumetric bone change will be calculated at 1 mm, 3 mm, and 5 mm apical to the alveolar crest using cross-sectional slices and 3D analysis software (Geomagic Control X).
  Data will be reported as mean change (mm for height; mm³ for volume) and standard deviation per group.
Soft Tissue Change from Baseline to 4 Months Using Intraoral Scans | Over the course of the study (4 months, From the time of study enrollment Alveolar Ridge Preservation [Visit 2] to 6-month dental implant placement [Visit 9]).
  Buccal soft tissue thickness will be evaluated using superimposed STL files obtained from intraoral digital scans. Scans will be collected at baseline, immediate post-surgery and 4 month post-surgery. Thickness will be measured at the mid-buccal point of the site, and changes will be reported as mean (mm) per group.

CONTACTS AND LOCATIONS:
Overall Officials: Hanae Saito, DDS MS CCRC, Principal Investigator — University of Maryland School of Dentistry
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No